CLINICAL TRIAL: NCT01015768
Title: Corneal Staining and Physiological Compromise After Eight Hours of Soft Contact Lens Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Responsible Party: Principal Investigator, Jerry R. Paugh, OD, PhD, Professor, Associate Dean or Research, Southern California College of Optometry at Marshall B. Ketchum University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 08-10
Record Dates: First submitted 2009-11-16; First posted 2009-11-18 (Estimated); Results first posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-08

CONDITIONS: Contact Lens-induced Corneal Fluorescein Staining
Keywords: corneal staining; barrier function; contact lenses; contact lens care solutions; contact lens material and care solution bioincompatibility

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test eye (Experimental): Uses ReNu Multiplus as multipurpose soaking solution
  Interventions: Device: ReNu Multiplus multipurpose disinfecting solution
- Control (Active Comparator): A new lens (PureVision) is soaked for 2 hours in non-preserved saline
  Interventions: Device: Control

INTERVENTIONS:
Device: ReNu Multiplus multipurpose disinfecting solution — A new lens (PureVision) soaked 6 hours to overnight in ReNu Multiplus
  Arms: Test eye
Device: Control — A new lens (PureVision) is soaked for two hours in non-preserved saline
  Arms: Control

SUMMARY:
The purpose of this study is to assess corneal staining and to measure the relative corneal epithelial "barrier" function (the degree to which the cornea can prevent penetration of colored sodium fluorescein dye into the eye) after 8 hours of wear with a known soft contact lens and multipurpose lens care solution combination.

DETAILED DESCRIPTION:
This investigation will evaluate corneal staining and epithelial barrier function after eight hours of contact lens wear, which is past the peak staining time and more typical of daily lens wear time. A silicone hydrogel lens and multipurpose solution combination shown to induce significant corneal staining ( e.g. equivalent Grade 3 out of Grade 4 scale) will be used to evaluate potential corneal compromise. The study will be a prospective, single-center, double-masked, contralateral, daily wear investigation in adapted soft contact lens wearers. After a three day washout period (without lens wear, lenses will then be worn on one day for eight hours. Corneal staining and barrier function will be determined for a regimen and a saline control situation for each subject. Staining will be graded using the Efron Grading Scale, and permeability data will be estimated as the fluorescein penetration rate, Pdc in nm/sec for the test and control condition.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Understand your rights as a research subject and give written informed consent by signing the Informed Consent Form, Subject Bill of Rights, and Patient Authorization for Use and Release of Health and Research Study Information (HIPAA form).
* Be likely to finish the entire study, understand the study instructions, and be willing to follow the instructions.
* Contact lens prescription between +4.00 D to -9.00 D (spherical equivalent).
* Best correctable visual acuity of at least 20/40 in each eye.
* Willing to de-adapt (do not wear) from habitual contact lenses for a period of at least two days prior to eligibility visit and at least two days prior to the testing day.
* Possess a functional spectacle (eyeglass) prescription to allow adequate vision during the de-adaptation and barrier function determination periods.
* No known allergies, which may interfere with contact lens wear.
* No known systemic (pertaining to general health) disease, or need for medication that may interfere with contact lens wear (i.e. antihistamines, beta-blockers, steroids).

Exclusion Criteria:

* Less than one month successful, full time (defined as at least 8 hours per day, and more than 5 days per week) soft lens wear.
* Clinically significant corneal swelling (greater than grade 3 or 4 on a 0-4 scale), corneal blood vessel growth (vascularization), corneal staining, bulbar redness, tarsal redness, or any other abnormality of the cornea that may cause unsafe contact lens wear.
* Any active ocular infection.
* Prior corneal refractive surgery (i.e., LASIK, PRK, etc).
* Have used medications within 24 hours of study entry or have an ongoing need to use ocular medication.
* Are taking part in any other study or have taken part in a study within the last 14 days
* Have a medical condition that your study eye doctor thinks may make it not appropriate for you to participate in this study.
* Are pregnant, or anticipate becoming pregnant during the course of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Paugh, OD, PhD, Study Director — Southern California College of Optometry at Marshall B. Ketchum University
Locations (1):
- Southern California Colege of Optometry, Fullerton, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eyes were randomized to one of two conditions.
Units Other Than Participants: eyes
Groups:
- Test Eye: A new PureVision contact lens is soaked in ReNu Multiplus disinfecting solution and worn for 8 hours
- Control: A new PureVision contact lens is soaked in non-preserved saline and worn for 8 hours
Period: Overall Study
Arm/Group | Test Eye | Control
Started | 30; 30 eyes | 30; 30 eyes
Completed | 26; 26 eyes | 26; 26 eyes
Not Completed | 4; 4 eyes | 4; 4 eyes
Not completed — Some subject data unuseable | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- All Participants: A new lens (PureVision) is soaked in ReNu Multiplus multipurpose soaking solution
  A new lens (PureVision) is soaked for 2 hours in non-preserved saline
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.2 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 30
Permeability Rate, Pdc [Mean (Standard Deviation); unit: nanometers per second] — Diffusion rate in nanometers per second
  nanometers per second | 0.05749 (0.038)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure Will be Corneal Epithelial Dye Diffusion Rate in Nanometers Per Second, for the Test and Control Eyes.
Description: The fluorescein dye diffusion rate in nanometers per second, is a diffusion rate into the corneal tissue. The fluorescein dye diffuses from the tears, where it is in high concentration, into the cornea, where it is in low concentration. It's diffusion is limited (or not) by the barrier properties and health of the epithelium.
Time Frame: After eight hours of wear
Population: Analysis was per protocol.
Measure: Mean (Standard Deviation); unit: nanometers per second
Units Other Than Participants: eyes
Groups:
- PHMB-containing Disinfectant: New lens soaked in B&L ReNu Multiplus disinfecting solution.
- Non-preserved Saline: New lens soaked for two hours in non-preserved saline
Arm/Group | PHMB-containing Disinfectant | Non-preserved Saline
Number analyzed (Participants) | 26 | 26
Number analyzed (eyes) | 26 | 26
nanometers per second | 0.0567 (0.039) | 0.0583 (0.038)

2. Primary Outcome: Permeability Rate, nm/Sec
Description: A penetration rate, in nm/sec
Time Frame: After eight hours of wear
Measure: Mean (Standard Deviation); unit: nm/sec
Units Other Than Participants: eyes
Arm/Group | Test Eye | Control
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 30 | 30
nm/sec | 0.057 (0.04) | 0.058 (0.04)

3. Secondary Outcome: The Secondary Outcome Measure Will be the Corneal Staining Grade, Compared Between the Test and Control Eye, as Well as Between the Baseline and Final Staining for Each Eye.
Description: Corneal staining represents corneal abrasion or damage. It is graded by us on a 0 - 4 scale (4 being worst) in five corneal sectors. The total score per cornea or eye is thus graded on a 0 - 20 total scale.
Time Frame: After eight hours of wear
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | PHMB-containing Disinfectant | Non-preserved Saline
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 30 | 30
score on a scale | 4.95 (2.4) | 4.52 (2.2)

ADVERSE EVENTS:
Arm/Group | Test Eye | Control
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
No limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes